CLINICAL TRIAL: NCT04953273
Title: Effectiveness of a Case Management Algorithm on Clinical Outcome After Consultations Requested in a Clinical Forensic Medicine Unit by Female Victims of Violence
Brief Title: A Case Management Algorithm for Women Victims of Violence
Acronym: VIGITRAUMA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2020_ 01; 2020-A02591-38 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2021-06-04; First posted 2021-07-07 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2022-04

CONDITIONS: Post-Traumatic Stress Disorder; Violence-Related Symptom
Keywords: Post-Traumatic Stress Disorder; Women Health; Physical Abuse; Forensic Medicine; Case-Management Algorithm
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vigitrauma (Experimental): Contact by phone at 3 weeks after the consultation in a clinical forensic medicine unit, and a second phone call if necessary.
  If the subject is not contacted after the second phone call, he will receive a postcard.
  Interventions: Other: Vigitrauma
- Control group (No Intervention): Usual follow-up.

INTERVENTIONS:
Other: Vigitrauma — Case management algorithm using early phone contact
  Arms: Vigitrauma

SUMMARY:
A considerable body of research has demonstrated that women who are victims of interpersonal violence are at substantially elevated risk for the development of post-traumatic stress disorder (PTSD). In France, victims can request a medico-legal examination in a clinical forensic medicine unit. Although these units are also a place for initial psychological examination, women often don't attend future scheduled appointments. Decision-making algorithm using phone contact are effective in suicide prevention. Our aim is to assess the effectiveness of case management algorithm using early phone contact compared to a control group treated as usual on clinical outcome after consultation requested in a clinical forensic medicine unit by female victims of violence.

Method: Prospective, multicenter, open-label, randomized controlled clinical trial, for women victims of violence. Victims randomized in VIGITRAUMA group will be contacted by phone at 3 weeks after the consultation in a clinical forensic medicine unit, and a second phone call can be done. If the subject is not contacted after the second phone call, he will receive a postcard.

Control group will benefit from usual follow-up.

All the subjects included will be then evaluated at 3 months, 6 months and 1 year during a phone call.

ELIGIBILITY:
Inclusion Criteria:

* Women
* 18 years and older
* Consultation requested in a clinical forensic medicine unit after being victim of violence
* The person was exposed to: death, threatened death, actual or threatened serious injury, or actual or threatened sexual violence (PTSD criterion A - DSM -5)
* With social insurance
* Consent to participate to the study

Exclusion Criteria:

* Do no consent to participate to the study
* Intrafamilial or intimate partner violence
* Do not speak french

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 756 (Estimated)
Dates: Start 2021-07-06 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Clinical Outcome | 3 months
  Rate of patients with a Clinical Global Impression (CGI) severity scale < 4
Clinical Outcome | 6 months
  Rate of patients with a Clinical Global Impression (CGI) severity scale < 4
Clinical Outcome | 12 months
  Rate of patients with a Clinical Global Impression (CGI) severity scale < 4

SECONDARY OUTCOMES:
Severity of post-traumatic stress disorder symptoms | 3 months, 6 months and 12 months
  Post-traumatic stress disorder Checklist Scale-5
General psychopathology | 3 months, 6 months and 12 months
  French version of Mini International Neuropsychiatric Interview (DSM 5)
Severity of somatic symptoms | 3 months, 6 months and 12 months
  Physical Health Questionnaire (PHQ-15)
Medical cost | 12 months
  Nnumber of hospitalizations, consultations, and drugs consummation
Judicial outcome | 12 months
  Number of days of temporary inability to work
Suicidal ideation intensity | 12 months
  The Beck Scale for Suicide Ideation (SSI) The Scale for Suicide Ideation (SSI; Beck, et al., 1979) is a brief 21-item scale that assesses the person's current intensity of attitudes, plans, and behaviors to commit suicide.
Number of suicide attempters | 12 months
  Suicide risk

CONTACTS AND LOCATIONS:
Overall Officials: Arnaud Leroy, MD, Principal Investigator — University Hospital, Lille
Locations (8):
- France (8):
  - University Hospital, Amiens, Amiens
  - General Hospital, Boulogne sur Mer, Boulogne-sur-Mer
  - University Hospital, Caen, Caen
  - General Hospital, Creil, Creil
  - University Hospital, Lille, Lille
  - University Hospital, Rouen, Rouen
  - General Hospital, Saint-Quentin, Saint-Quentin
  - General Hospital, Valenciennes, Valenciennes